CLINICAL TRIAL: NCT05122806
Title: Biological Characterization of Advanced ALK-rearranged Non-small Cell Lung (NSCLC) Cancer Included in EXPLOREALK Study
Brief Title: Analysis of Biological Characteristics of Advanced ALK-rearranged NSCLC
Acronym: BIOEXALK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GroupeFDPC; GFPC 08-2020 (Other: GroupeFDPC)
Record Dates: First submitted 2021-09-06; First posted 2021-11-17 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer; ALK Gene Rearrangement Positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Base Sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bioexalk cohort (Other): All patients included in Explore ALK GFPC 03-2019 study who agree to participate in Bioexalk.
  Interventions: Genetic: RNAseq

INTERVENTIONS:
Genetic: RNAseq — 1. Tissue : RNAseq will be performed on tumor biopsy (10 slides of 5 microns) to identify the ALK fusion partner and its variant and associated co-mutations.
  2. ctDNA : NGS panel on DNA including a large panel of fusions and mutations will be performed on blood samples
  Other Names: DNA NGS

SUMMARY:
BioEXALK is a prospective study evaluating the biological characteristics of advanced ALK-rearranged NSCLC treated with next generation TKIs in first line, included in the national EXPLORE ALK cohort (GFPC 03-2019), a non-interventional, national, multi-center cohort of ALK-rearranged NSCLC patients.

BioExALK study will be proposed to every patient included in the Explore ALK GFPC 03-2019 study.

Biological analysis will be performed on tumor tissue at diagnosis and at the time of disease progression when available and on circulating tumor DNA (ctDNA).

For plasma testing, after obtained patient consent, blood samples will be taken and analyzed at the Léon Bérard Center (Lyon).

Biological analysis on tissue obtained at diagnosis and at disease progression will be collected and be sent for centralized analysis to the Rouen University Hospital.

DETAILED DESCRIPTION:
BioEXALK is a prospective study evaluating the biological characteristics of advanced ALK-rearranged NSCLC treated with new generation TKIs in first line, included in the national EXPLORE ALK cohort (GFPC 03-2019).

Explore ALK GFPC 03-2019 is a non-interventional, national, multi-center cohort of ALK-rearranged NSCLC patients, whose RCB reference is 2020-A00771-38 and which obtained an approval from the IDF II Ethic Committee on 25/05/2020. Biological analysis will be performed on tissue at diagnosis and at the time of disease progression when available and on circulating tumor DNA (ctDNA) on three timepoints (diagnosis, at first tumor evaluation and at the time of disease progression).

* Tissue : RNAseq will be performed on tumor biopsy (10 slides of 5 microns) to identify the ALK fusion partner and its variant and associated co-mutations..
* ctDNA : NGS panel on DNA including a large panel of fusions and mutations will be performed on blood samples (30mL on EDTA or STRECKs tubes) at diagnosis, at the time of the first evaluation and at the time of progression).

For plasma testing, after obtained patient consent, blood samples (35mL on EDTA or STRECKs tubes) at diagnosis, at the first evaluation and at disease progression will be taken.

The ALKis include alectinib and brigatinib as first-line therapy or other drugs with marketing authorizations (lorlatinib, entrectinib) or in early access programs (EAPs).

Liquid biopsies will be analyzed with a NGS panel allowing the identification of ALK fusion partners and resistance mechanisms (mutations, fusions, copy number variations). Samples will be sent for centralized analysis to the Léon Bérard Center (Lyon).

For biological analysis on tissue obtained at diagnosis, the ALK fusion partner and its variant will be identified by RNAseq. Whenever a tissue re-biopsy is performed at the time of disease progression as part of the standard of care management of the patient, the remaining tissue sample will be collected as part of the BioExALK study, so that RNAseq analysis will be performed to look for resistance mechanisms. Tissue samples (10 slides of 5 microns) will be sent for centralized analysis to the Rouen University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB/IV NSCLC non eligible to locoregional treatment with curative intent
* ALK rearrangement confirmed by IHC and/or FISH or NGS according to local methods
* Patient included in the EXPLORE ALK study
* Age > or = 18 years
* Patient treated with first-line new generation ALKi
* Patient agrees to sign an informed consent form and to collect blood samples at inclusion, first tumor evaluation and progression and for whom tumor biopsy at diagnosis is available
* Patient enrolled in the french National Health Insurance program or with a third- party payer

Exclusion Criteria:

* Patients who do not wish to participate in Bioexalk
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of treatment initiation up to 72 months
  PFS assessed by local review using RECIST v1.1, defined as time from treatment initiation to the first clinical or radiological progression or death from any cause

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of treatment initiation up to 72 months
  OS defined as time from treatment initiation to death from any cause.
Duration of Response (DoR) | From date of treatment initiation up to 72 months
  DoR assessed by local review using RECIST v1.1, defined as time from treatment initiation to the first clinical or radiological progression, death, consent withdrawn, adverse event, protocol deviations, lost to follow-up, or initiation of a new line of anticancer therapy.
Overall Response Rate (ORR) | From date of treatment initiation up to 72 months
  ORR defined as objective response rate of complete response or partial response measured by local review RECIST v1.1.
Circulating tumoral DNA (ctDNA) clearance on Progression Free Survival (PFS) of stage IV ALK-rearranged NSCLC patients | From date of treatment initiation up to 72 months
  ctDNA clearance will be determine as clearance of the fusion when detectable and/or clearance of relevant mutations when fusion not detected
Circulating tumoral DNA (ctDNA) clearance on Overall Survival (OS) of stage IV ALK-rearranged NSCLC patients | From date of treatment initiation up to 72 months
  ctDNA clearance will be determine as clearance of the fusion when detectable and/or clearance of relevant mutations when fusion not detected
Circulating tumoral DNA (ctDNA) clearance on Duration of Response (DoR) of stage IV ALK-rearranged NSCLC patients | From date of treatment initiation up to 72 months
  ctDNA clearance will be determine as clearance of the fusion when detectable and/or clearance of relevant mutations when fusion not detected
Circulating tumoral DNA (ctDNA) clearance on Overall Response Rate (ORR) of stage IV ALK-rearranged NSCLC patients | From date of treatment initiation up to 72 months
  ctDNA clearance will be determine as clearance of the fusion when detectable and/or clearance of relevant mutations when fusion not detected
Description of mechanisms of resistance associated with first-line tyrosine kinase inhibitors | From date of treatment initiation up to 72 months
  The following mechanisms of resistance will be assessed: secondary mutations on ALK, mutations or translocations on other genes of interest, histological transformations
Description of mechanism of resistance associated with each ALK-fusion partner | From date of treatment initiation up to 72 months
  The following mechanisms of resistance will be assessed: secondary mutations on ALK, mutations or translocations on other genes of interest, histological transformations
Concordance between ALK fusion partner and co-mutations | From date of treatment initiation up to 72 months
  ALK fusion partner and co-mutation identifications based on liquid and tissue biopsies at Baseline
Impact of presence or absence of serum Anti-ALK antibodies at diagnosis on OS | From date of treatment initiation up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Christos CHOUAID, Study Director — Groupe Francais De Pneumo-Cancerologie
Locations (46):
- France (46):
  - Pneumologie CHU Félix Guyon, Saint-Denis, La Réunion
  - Centre Hospitalier d'Aix en Provence, Aix-en-Provence
  - Pneumologie CHU, Amiens
  - Centre Hospitalier Universitaire, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospitalier du Morvan, Brest
  - Centre François Baclesse, Caen
  - Pneumologie CH Métropole Savoie, Chambéry
  - Oncologie CLCC Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Pneumologie CH Eure-Seine, Évreux
  - Pneumologie CHD Vendée, La Roche-sur-Yon
  - Pneumologie Hôpital Mignot, Le Chesnay
  - Pneumologie CH, Le Mans
  - Oncologie Centre Oscar Lombret, Lille
  - Pneumologie Hôpital Calmette, Lille
  - Pneumologie CHU Limoges, Limoges
  - Hôpital du Scorff, Lorient
  - Pneumologie Hôpital privé Jean Mermoz, Lyon
  - Centre Léon Bérard, Lyon
  - Oncologie Hôpital François Quesnay, Mantes-la-Jolie
  - Pneumologie Hôpital Européen, Marseille
  - Oncologie Institut Paoli Calmette, Marseille
  - Hôpital Nord, Marseille
  - Hôpital de Meaux, Meaux
  - Oncologie Institut du Cancer de Montpellier, Montpellier
  - Oncologie CH Morlaix, Morlaix
  - Pneumologie CHR, Orléans
  - Oncologie Institut Curie, Paris
  - Pneumologie Centre Hospitalier, Pau
  - Hôpital du Haut Leveque, Pessac
  - CHU Pontchailloux, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Pneumologie Hôpital Yves Le Foll, Saint-Brieuc
  - CHU La Réunion Site Sud, Saint-Pierre
  - Institut Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Pneumologie Hôpital Foch, Suresnes
  - Pneumologie HIA, Talence
  - Pneumologie Hôpital Sainte Musse, Toulon
  - Hôpital d'Instruction des Armées Ste Anne, Toulon
  - Hôpital Larrey, Toulouse
  - Oncologie CH Bretagne-Atlantique, Vannes
  - Centre Hospitalier de Villefranche sur Saone, Villefranche-sur-Saône
  - Oncologie Institut Gustave Roussy, Villejuif
  - Pneumologie CHI, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No